CLINICAL TRIAL: NCT01631357
Title: Phase II/III Study of Chemotherapy Combination With Autologous Cytokine-Induced Killer Cell Immunotherapy in Stage IIIb-IV Squamous Non-Small-Cell Lung Cancer
Brief Title: Study of Chemotherapy Combination With Autologous Cytokine-Induced Killer Cell Immunotherapy to Treat Lung Cancer
Acronym: CIK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIH-RXB-201205001
Record Dates: First submitted 2012-05-27; First posted 2012-06-29 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2014-11

CONDITIONS: Non-small Cell Lung Cancer; Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: CIK+CT (Experimental): Arm 1: We design chemotherapy combination with CIK cell immunotherapy as a experimential arm.
  Interventions: Biological: CIK cell; Drug: Gemcitabine Injection; Drug: Cisplatin injection
- Arm 2: CT (Active Comparator): Arm 2: We design chemotherapy alone as a control arm
  Interventions: Drug: Gemcitabine Injection; Drug: Cisplatin injection

INTERVENTIONS:
Biological: CIK cell — CIK cell injection
  Other Names: Cytokine-induced killer cell
  Arms: Arm 1: CIK+CT
Drug: Gemcitabine Injection — Gemcitabine injection
  Other Names: Gemcitabine
Drug: Cisplatin injection — Cisplatin injection
  Other Names: Cisplatin

SUMMARY:
This randomized, multicenter,open-label phase II/III study is to evaluate the effects of chemotherapy combination with autologous cytokine-induced killer Cell immunotherapy in patients with stage IIIb-IV squamous non-small-cell lung cancer

DETAILED DESCRIPTION:
1. Phase II/III study,
2. Randomized, multicenter, open-label study,
3. Evaluated the effects of chemotherapy combination with autologous cytokine-induced killer Cell immunotherapy compared with chemotherapy in patients with stage IIIb-IV squamous non-small-cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Sex: male or female
* Age: from 18 to 80 years
* Histology: squamous non-small-cell lung cancer
* Clinical stage: from stage IIIb to stage IV
* Therapy: not received chemotherapy, radiotherapy, or immunotherapy before entry into this study
* Karnofsky performance status: more than 50%
* Expected survival: more than 2 months
* Laboratory tests results 7 days before the start of treatment:

White blood cells: more than 3.0 × 109/L Platelets: more than 100 × 109/L Neutrophils: more than 1.5 × 109/L Hemoglobin: more than 80g/L Serum glutamate pyruvate transaminase: less than 2.5 folds of the upper normal limit (ULN) Serum glutamic-oxal (o) acetic transaminase: less than 2.5 × ULN Serum bilirubin: less than 1.25 × ULN Serum creatinine: less than 1.25 × ULN

* pregnancy test: the test of women of child-bearing period must be negative 7 days before the start of treatment
* Contraception: male and female subjects of child-bearing period must adopt a reliable method of contraception before entry into this study until 30 days after stopping this study
* Informed consent: subject must have the ability to understand and voluntarily sign a written informed consent

Exclusion Criteria:

* History of neoplasms: other neoplasms
* Medical history: mental disease, or congestive heart failure, or severe coronary artery disease, or cardiac arrhythmias, or concomitant corticosteroid therapy
* History of allergies: allergic to the study drugs
* Metastasis: clinical symptoms of brain metastasis
* Other clinical trial: the subject received other clinical trial before this study
* Laboratory tests: the serum test of human immunodeficiency virus, or hepatitis B virus, or hepatitis C virus was positive
* Woman: pregnant or lactating women
* Compliance: poor compliance
* History of neoplasms: other neoplasms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | up to 3 years
  PFS was measured from the date of randomization to the first disease progression or to death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | up to 3 years
  OS was measured from the date of randomization until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiubao Ren, MD, PhD, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China